CLINICAL TRIAL: NCT01059435
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 785 in Healthy Men and Postmenopausal Women
Brief Title: A First-in-human Study Evaluating Romosozumab (AMG 785) in Healthy Men and Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20060220
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Osteopenia
Keywords: Amgen; First in Human; Postmenopausal; Phase 1
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Participants were randomized to receive a single dose of matching placebo administered by subcutaneous or intravenous injection.
  Interventions: Drug: Placebo
- Romosozumab (Experimental): Participants were randomized to receive a single dose of romosozumab administered by subcutaneous or intravenous injection. The starting dose was 0.1 mg/kg, with sequential escalation up to 10 mg/kg.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered subcutaneously or intravenously
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab
Drug: Placebo — Administered subcutaneously or intravenously
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of romosozumab following single dose subcutaneous (SC) or intravenous (IV) administration in healthy men and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or female between 45 to 59 years of age, inclusive
* Postmenopausal females defined as 12 continuous months of spontaneous amenorrhea confirmed by a serum follicle-stimulating hormone (FSH) result > 40mIU/mL, or 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy)
* Males must agree to use a condom during sexual intercourse with female partners who are of reproductive potential and to have their female partners use an additional effective means of contraception or to abstain from sexual intercourse for the duration of the study
* Has no history or evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Exclusion Criteria:

* Diagnosed with any condition that will affect bone metabolism
* Administration of the following medications within 6 months before study drug administration:
* Hormone replacement therapy [Infrequent use of estrogen vaginal creams (< 3 times per week) is allowed.]
* Calcitonin
* Parathyroid hormone (or any derivative)
* Supplemental Vitamin D > 1,000 IU/day
* Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the enrollment date are allowed)
* Anabolic steroids
* Calcitriol, and available analogues
* Administration of the following medications within 12 months before study drug administration:
* Bisphosphonates
* Fluoride for osteoporosis
* Administration of herbal medications within 2 weeks or 5 half-lives (whichever is longer) before study drug administration
* Greatly differing levels of physical activity or constant levels of intense physical exercise during the 6 months before study drug administration
* Routine alcohol intake of > 2 drinks per day, on average, within 6 months of study drug administration
* Known sensitivity to mammalian-derived drug preparations
* Known to be hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus (HIV) positive, or a known diagnosis of acquired immunodeficiency syndrome (AIDS)
* Any organic or psychiatric disorder which may pose a risk to subject safety and may prevent the subject from completing the study or interfere with the interpretation of the study results
* Unavailable for follow-up assessment or any concerns for subject's compliance with the protocol procedures
* Any other condition that might reduce the chance of obtaining data required by the protocol or that might compromise the ability to give truly informed consent
* Has a history of drug or alcohol abuse with the last 12 months and/or a positive urine test result at screening or admission
* Has any clinically significant abnormality during the screening physical examination, electrocardiogram (ECG), or laboratory evaluation
* Has participated in another clinical study within 4 weeks of screening or within 5 times the half-life of the investigational agent in the other clinical study, if known
* Weight ≥ 98 kilograms (216 pounds) and/or height ≥ 78 inches
* Has donated or lost 400 milliliters or more of blood or plasma within 8 weeks of study drug administration

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2006-12-13 (Actual); Primary Completion 2007-07-06 (Actual); Study Completion 2007-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Padhi D, Jang G, Stouch B, Fang L, Posvar E. Single-dose, placebo-controlled, randomized study of AMG 785, a sclerostin monoclonal antibody. J Bone Miner Res. 2011 Jan;26(1):19-26. doi: 10.1002/jbmr.173. PMID 20593411
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center study conducted in the USA. The first participant enrolled on 13 December 2006 and the last participant completed the study on 06 July 2007.
Pre-assignment Details: Participants were enrolled sequentially into 1 of 6 dose cohorts. Healthy postmenopausal women were randomized to romosozumab or placebo in a 3:1 ratio at 0.1, 0.3, 1 mg/kg SC, 1 mg/kg IV, 3, 5 mg/kg SC, 10 mg/kg SC, or 10 mg/kg IV; healthy men received romosozumab SC or IV, placebo SC or IV in a 3:3:1:1 ratio at doses of 1 mg/kg or 10 mg/kg.
Groups:
- Placebo SC: Participants received a single subcutaneous (SC) injection of matching placebo.
- Romosozumab 0.1 mg/kg SC: Participants received a single subcutaneous injection of 0.1 mg/kg romosozumab.
- Romosozumab 0.3 mg/kg SC: Participants received a single subcutaneous injection of 0.3 mg/kg romosozumab.
- Romosozumab 1.0 mg/kg SC: Participants received a single subcutaneous injection of 1.0 mg/kg romosozumab.
- Romosozumab 3.0 mg/kg SC: Participants received a single subcutaneous injection of 3.0 mg/kg romosozumab.
- Romosozumab 5.0 mg/kg SC: Participants received a single subcutaneous injection of 5.0 mg/kg romosozumab.
- Romosozumab 10.0 mg/kg SC: Participants received a single subcutaneous injection of 10.0 mg/kg romosozumab.
- Placebo IV: Participants received a single intravenous (IV) injection of matching placebo.
- Romosozumab 1.0 mg/kg IV: Participants received a single intravenous injection of 1.0 mg/kg romosozumab.
- Romosozumab 5.0 mg/kg IV: Participants received a single intravenous injection of 5.0 mg/kg romosozumab
Period: Overall Study
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Started | 14 | 6 | 8 | 9 | 6 | 9 | 6 | 4 | 6 | 6
Received Study Drug | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
Completed | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV | Total
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6 | 72
Age, Continuous [Mean (Standard Deviation); unit: years]
  SC Dosing | 52.79 (4.17) | 53.00 (3.95) | 53.33 (3.20) | 52.00 (4.64) | 55.00 (4.05) | 51.89 (2.32) | 52.50 (4.32) | NA (NA) — SC dosing cohorts are reported in this row | NA (NA) — SC dosing cohorts are reported in this row | NA (NA) — SC dosing cohorts are reported in this row | 52.80 (3.79)
  IV Dosing | NA (NA) — IV dosing cohorts are reported in this row | NA (NA) — IV dosing cohorts are reported in this row | NA (NA) — IV dosing cohorts are reported in this row | NA (NA) — IV dosing cohorts are reported in this row | NA (NA) — IV dosing cohorts are reported in this row | NA (NA) — IV dosing cohorts are reported in this row | NA (NA) — IV dosing cohorts are reported in this row | 52.50 (4.43) | 49.33 (4.63) | 51.00 (3.35) | 50.75 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 3 | 3 | 56
  Male | 2 | 0 | 0 | 3 | 0 | 3 | 0 | 2 | 3 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 6
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hispanic or Latino | 12 | 6 | 6 | 9 | 6 | 9 | 5 | 2 | 4 | 6 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Serious adverse events were any events that were fatal, were life-threatening (placed the participant at immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, were congenital anomalies or birth defects, or were other significant medical hazards.
  Relatedness to investigational product was assessed by the investigator by means of the question: "Is there a reasonable possibility that the event may have been caused by the investigational product?'
Time Frame: Adverse events were collected from the first dose of treatment up until day 29 for the 0.1 mg/kg and 0.3 mg/kg SC treatment groups, up to 57 days for the 1 mg/kg and 3 mg/kg IV/SC groups and for up to 85 days for the 5 mg/kg and 10 mg/kg SC/IV groups.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
Participants
  Any adverse event | 9 | 4 | 4 | 1 | 5 | 6 | 5 | 2 | 1 | 2
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Treatment-related adverse events | 5 | 4 | 2 | 0 | 3 | 4 | 5 | 0 | 1 | 1
  Serious treatment-related adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Discontinuations due to adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Developed Anti-romosozumab Antibodies
Description: Binding anti-romosozumab antibody titers were assessed using a validated electrochemiluninescence (ECL) immunoassay. The limit of detection for this assay was 3.91 ng/mL of anti-romosozumab antibody in neat serum. Samples found to be positive for binding antibodies were further tested using a validated bioassay to determine if the antibodies were able to neutralize the activity of romosozumab. The limit of detection for this assay was ≥ 0.75 μg/mL.
Time Frame: Day 29 (all participants), day 57 (1, 3, 5, and 10 mg/kg treatment groups only) and at day 85 (5 and 10 mg/kg teatment groups only).
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
participants
  Binding antibody positive | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2
  Neutralizing antibody positive | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Romosozumab
Time Frame: Predose up to day 29 for participants receiving 0.1 or 0.3 mg/kg romosozumab, up to day 57 for participants receiving 1 or 3 mg/kg romosozumab, and up to day 85 for participants receiving 5 or 10 mg/kg romosozumab.
Population: All treated participants who received subcutaneous romosozumab
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6
ng/mL | 375 (182) | 1280 (653) | 4890 (1780) | 21300 (5170) | 33500 (8290) | 75200 (15900)

4. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Romosozumab
Time Frame: as for outcome 3
Population: All treated participants who received subcutaneous romosozumab
Measure: Median (Full Range); unit: days
Arm/Group | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6
days | 1.5 [0.5 to 7] | 2.5 [2 to 5] | 3 [2 to 14] | 5 [4 to 7] | 5 [3 to 7] | 4.5 [2 to 7]

5. Secondary Outcome: Initial Concentration Following IV Administration (C0) of Romosozumab
Time Frame: Day 1 at the end of infusion
Population: All treated participants who received intravenously administered romosozumab
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 6 | 6
ng/mL | 24900 (4670) | 132000 (13700)

6. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity for Romosozumab
Time Frame: as for outcome 3
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 6
µg*hr/mL | 78.5 (22.6) | 288 (144) | 1480 (605) | 8170 (1810) | 16900 (4350) | 43400 (8550) | 3020 (989) | 24400 (4400)

7. Secondary Outcome: Apparent Clearance (CL/F) / Clearance (CL) for Romosozumab
Time Frame: as for outcome 3
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 6
mL/hr/kg | 1.39 (0.489) | 1.35 (0.841) | 0.873 (0.647) | 0.383 (0.0901) | 0.319 (0.0998) | 0.236 (0.0370) | 0.362 (0.117) | 0.210 (0.0361)

8. Secondary Outcome: Half-life Associated With the Beta (Plateau) Phase of Elimination for Romosozumab
Description: The plateau (beta, β) phase half-life (t½,β) was calculated from the natural log of 2 divided by the beta phase rate constant (λβ). λβ for a subject was estimated by linear regression of at least 3 contiguous time points that followed the Cmax and constituted a distinct phase that preceded the terminal phase.
Time Frame: as for outcome 3
Population: All treated participants who received 3, 5, or 10 mg/kg romosozumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 9 | 6 | 0 | 6
days |  |  |  | 11.1 (3.70) | 12.9 (3.14) | 18.0 (3.54) |  | 10.6 (1.70)

9. Secondary Outcome: Half-life Associated With the Gamma (Terminal) Phase of Elimination for Romosozumab
Description: The terminal (gamma, γ) phase half-life (t½,γ) was calculated from the natural log of 2 divided by the terminal rate constant (λz).
Time Frame: as for outcome 3
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 9 | 6 | 6 | 6
days | 5.20 (1.36) | 5.13 (0.640) | 5.50 (0.322) | 6.68 (0.961) | 5.81 (0.874) | 5.88 (1.60) | 4.49 (0.974) | 4.93 (0.639)

10. Secondary Outcome: Maximum Effect for Serum Type 1 Aminoterminal Propeptide (P1NP)
Description: Defined as the maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
ng/mL | 69.8 (32.0) | 57.7 (22.8) | 60.9 (14.4) | 60.7 (10.8) | 100.8 (49.6) | 125.1 (44.2) | 141.4 (24.8) | 77.0 (35.3) | 76.3 (19.8) | 173.4 (43.3)

11. Secondary Outcome: Time to Maximum Effect of P1NP
Description: Defined as the time to maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Median (Full Range); unit: days
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days | 39.5 [1.0 to 64.0] | 11.0 [6.0 to 29.0] | 4.5 [1.0 to 15.0] | 15.0 [11.0 to 57.0] | 22.0 [15.0 to 22.0] | 22.0 [15.0 to 29.0] | 25.5 [22.0 to 36.0] | 43.0 [1.0 to 57.0] | 15.0 [11.0 to 22.0] | 18.5 [15.0 to 29.0]

12. Secondary Outcome: Area Under the Curve From Day 0 to Day 29 (AUC0-29) for P1NP
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*ng/mL | 1529 (633) | 1431 (548) | 1564 (377) | 1473 (304) | 2300 (1099) | 2780 (1007) | 2986 (306) | 1714 (782) | 1794 (434) | 3940 (944)

13. Secondary Outcome: Area Under the Curve From Day 0 to the Last Sampling Time Point (AUC0-t) for P1NP
Time Frame: Predose up to day 29 for participants receiving 0.1 or 0.3 mg/kg romosozumab, up to day 57 for participants receiving 1 or 3 mg/kg romosozumab, and up to day 85 for participants receiving 5 or 10 mg/kg romosozumab,
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*ng/mL | 3234 (1462) | 1431 (548) | 1564 (377) | 2782 (513) | 3962 (1702) | 6759 (2434) | 7846 (1264) | 4487 (2352) | 3138 (723) | 8976 (2531)

14. Secondary Outcome: Maximum Effect for Serum C-telopeptide (sCTX)
Description: Defined as the minimum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
ng/mL | 0.3 (0.2) | 0.4 (0.2) | 0.3 (0.1) | 0.3 (0.1) | 0.4 (0.1) | 0.2 (0.1) | 0.2 (0.1) | 0.3 (0.2) | 0.2 (0.1) | 0.2 (0.1)

15. Secondary Outcome: Time to Maximum Effect of sCTX
Description: Defined as the time to minimum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Median (Full Range); unit: days
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days | 1.0 [1.0 to 36.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 43.0] | 1.0 [1.0 to 50.0] | 8.0 [1.0 to 78.0] | 6.0 [1.0 to 22.0] | 18.5 [1.0 to 43.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 64.0]

16. Secondary Outcome: Area Under the Curve From Day 0 to Day 29 (AUC0-29) for sCTX
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*ng/mL | 20 (8) | 21 (6) | 18 (5) | 15 (6) | 14 (3) | 11 (4) | 8 (3) | 21 (8) | 13 (3) | 12 (5)

17. Secondary Outcome: Area Under the Curve From Day 0 to the Last Sampling Time Point (AUC0-t) for sCTX
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*ng/mL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*ng/mL | 37 (18) | 21 (6) | 18 (5) | 30 (13) | 29 (7) | 41 (18) | 40 (15) | 44 (20) | 26 (6) | 44 (13)

18. Secondary Outcome: Maximum Effect for Osteocalcin
Description: Defined as the maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
µg/L | 28.9 (8.1) | 25.6 (8.0) | 25.8 (4.8) | 26.6 (5.5) | 36.9 (10.9) | 39.0 (12.7) | 53.9 (10.5) | 35.9 (13.9) | 28.8 (7.7) | 53.5 (12.8)

19. Secondary Outcome: Time to Maximum Effect of Osteocalcin
Description: Defined as the time to maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Median (Full Range); unit: days
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days | 29.0 [2.0 to 57.0] | 15.0 [2.0 to 15.0] | 18.5 [2.0 to 38.0] | 22.0 [11.0 to 36.0] | 22.0 [22.0 to 29.0] | 29.0 [29.0 to 50.0] | 36.0 [26.0 to 57.0] | 34.0 [5.0 to 64.0] | 22.0 [11.0 to 36.0] | 32.5 [29.0 to 43.0]

20. Secondary Outcome: Area Under the Curve From Day 0 to Day 29 (AUC0-29) for Osteocalcin
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*µg/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*µg/L | 617 (209) | 611 (191) | 658 (153) | 570 (139) | 753 (234) | 757 (225) | 881 (162) | 759 (286) | 559 (73) | 973 (212)

21. Secondary Outcome: Area Under the Curve From Day 0 to the Last Sampling Time Point (AUC0-t) for Osteocalcin
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*µg/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*µg/L | 1259 (505) | 611 (191) | 658 (153) | 1129 (256) | 1487 (453) | 2470 (827) | 2964 (563) | 1897 (519) | 1132 (131) | 2988 (460)

22. Secondary Outcome: Maximum Effect for Bone-specific Alkaline Phosphatase (BSAP)
Description: Defined as the maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
µg/L | 21.0 (5.7) | 18.0 (6.7) | 17.2 (3.2) | 17.7 (4.7) | 26.1 (7.8) | 24.6 (8.6) | 29.9 (8.2) | 19.6 (3.7) | 15.9 (4.5) | 36.4 (15.9)

23. Secondary Outcome: Time to Maximum Effect of BSAP
Description: Defined as the time to maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Median (Full Range); unit: days
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days | 36.0 [4.0 to 78.0] | 16.5 [4.0 to 29.0] | 13.0 [6.0 to 19.0] | 15.0 [8.0 to 29.0] | 22.0 [22.0 to 22.0] | 22.0 [22.0 to 36.0] | 22.0 [15.0 to 29.0] | 46.5 [6.0 to 85.0] | 13.5 [6.0 to 50.0] | 29.0 [22.0 to 36.0]

24. Secondary Outcome: Area Under the Curve From Day 0 to Day 29 (AUC0-29) for BSAP
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*µg/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*µg/L | 462 (157) | 460 (172) | 460 (127) | 422 (100) | 588 (152) | 540 (210) | 639 (176) | 448 (73) | 376 (102) | 780 (325)

25. Secondary Outcome: Area Under the Curve From Day 0 to the Last Sampling Time Point (AUC0-t) for BSAP
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*µg/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*µg/L | 958 (428) | 460 (172) | 460 (127) | 815 (190) | 1120 (303) | 1496 (527) | 1860 (508) | 1138 (191) | 731 (177) | 2033 (780)

26. Secondary Outcome: Maximum Effect for Intact Parathyroid Hormone (iPTH)
Description: Defined as the maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
ng/L | 43.3 (12.6) | 38.7 (11.9) | 54.5 (13.1) | 49.9 (20.5) | 62.8 (10.9) | 66.0 (20.0) | 76.3 (15.7) | 64.8 (27.8) | 52.7 (20.1) | 59.7 (14.9)

27. Secondary Outcome: Time to Maximum Effect of iPTH
Description: Defined as the time to maximum value postdose.
Time Frame: as for outcome 3
Population: All treated participants
Measure: Median (Full Range); unit: days
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days | 11.0 [1.0 to 71.0] | 11.0 [1.0 to 15.0] | 25.5 [15.0 to 29.0] | 22.0 [3.0 to 43.0] | 22.0 [1.0 to 29.0] | 22.0 [8.0 to 50.0] | 15.0 [1.0 to 50.0] | 25.5 [1.0 to 71.0] | 11.0 [1.0 to 57.0] | 18.5 [8.0 to 43.0]

28. Secondary Outcome: Area Under the Curve From Day 0 to Day 29 (AUC0-29) for iPTH
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*ng/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*ng/L | 817 (295) | 823 (202) | 1234 (341) | 1002 (405) | 1270 (198) | 1240 (342) | 1422 (411) | 1235 (488) | 1074 (406) | 1239 (267)

29. Secondary Outcome: Area Under the Curve From Day 0 to the Last Sampling Timepoint (AUC0-t) for iPTH
Time Frame: as for outcome 3
Population: All treated participants
Measure: Mean (Standard Deviation); unit: days*ng/L
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
days*ng/L | 1592 (689) | 823 (202) | 1234 (341) | 1971 (850) | 2523 (406) | 3483 (1057) | 4195 (1144) | 3100 (1077) | 2072 (749) | 3515 (1127)

30. Secondary Outcome: Percent Change From Baseline in Sclerostin
Time Frame: Baseline and days 15, 29, 43, 57, 71, and 85
Population: All treated participants; only participants who received ≥ 1 mg/kg romosozumab/placebo were assessed after day 29 and only participants who received 5 or 10 mg/kg romosozumab/placebo were assessed on days 71 and 85.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
percent change
  Day 15 | 53.2 (54.3) | 465.5 (49.9) | 835.1 (130.4) | 2123.8 (377.6) | 7965.9 (792.9) | 12375.7 (1375.4) | 17774.8 (2444.0) | 6.7 (11.4) | 3776.0 (461.5) | 14230.0 (2428.1)
  Day 29 | -8.4 (7.0) | 129.0 (33.3) | 183.0 (19.6) | 717.4 (92.4) | 5140.2 (373.7) | 9763.2 (1252.8) | 18870.9 (2707.3) | -4.3 (8.7) | 816.7 (222.3) | 11715.5 (2177.0)
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 43 | -9.8 (14.1) |  |  | 223.2 (18.1) | 1988.3 (339.9) | 4968.7 (714.7) | 13902.7 (2381.9) | 4.9 (8.7) | 196.1 (48.7) | 4576.0 (1086.7)
  Day 57: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 57 | -3.7 (8.6) |  |  | 83.4 (14.5) | 810.2 (169.9) | 2004.9 (421.5) | 6469.6 (1000.3) | 15.6 (0.6) | 49.9 (17.4) | 1430.0 (538.0)
  Day 71: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 71 | 86.9 (88.3) |  |  |  |  | 610.4 (151.6) | 2080.8 (689.0) | -5.5 (5.4) |  | 426.9 (119.6)
  Day 85: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 85 | 11.6 (16.6) |  |  |  |  | 232.1 (49.0) | 758.0 (270.1) | 0.8 (13.4) |  | 109.8 (30.6)

31. Secondary Outcome: Serum Calcium Over Time
Time Frame: Dday 1 predose and at 4, 6, 8, 10, and 12 hours, days 2, 3, 4, 5, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, and 85
Population: All treated participants; only participants who received ≥ 1 mg/kg romosozumab/placebo were assessed after day 29 and only participants who received 5 or 10 mg/kg romosozumab/placebo were assessed after day 57.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
mg/dL
  Day 1 Pre-dose | 9.49 (0.34) | 9.45 (0.38) | 9.50 (0.33) | 9.48 (0.27) | 9.42 (0.25) | 9.53 (0.26) | 9.38 (0.24) | 9.60 (0.22) | 9.23 (0.15) | 9.37 (0.15)
  Day 1 Hour 4 | 9.46 (0.30) | 9.62 (0.19) | 9.45 (0.26) | 9.38 (0.16) | 9.38 (0.15) | 9.59 (0.27) | 9.35 (0.40) | 9.45 (0.21) | 9.43 (0.22) | 9.40 (0.17)
  Day 1 Hour 6 | 9.49 (0.26) | 9.38 (0.22) | 9.50 (0.14) | 9.47 (0.17) | 9.60 (0.24) | 9.48 (0.35) | 9.25 (0.36) | 9.18 (0.13) | 9.38 (0.31) | 9.40 (0.15)
  Day 1 Hour 8 | 9.38 (0.22) | 9.47 (0.29) | 9.33 (0.23) | 9.29 (0.18) | 9.28 (0.12) | 9.42 (0.28) | 9.27 (0.33) | 9.38 (0.21) | 9.35 (0.10) | 9.22 (0.12)
  Day 1 Hour 10 | 9.53 (0.26) | 9.62 (0.31) | 9.50 (0.27) | 9.40 (0.30) | 9.38 (0.19) | 9.36 (0.31) | 9.28 (0.27) | 9.50 (0.22) | 9.45 (0.16) | 9.42 (0.15)
  Day 1 Hour 12 | 9.53 (0.28) | 9.55 (0.27) | 9.57 (0.31) | 9.49 (0.31) | 9.37 (0.34) | 9.52 (0.26) | 9.27 (0.34) | 9.40 (0.24) | 9.47 (0.19) | 9.45 (0.19)
  Day 2 | 9.46 (0.34) | 9.55 (0.21) | 9.23 (0.28) | 9.39 (0.21) | 9.37 (0.33) | 9.46 (0.29) | 9.23 (0.29) | 8.55 (1.77) | 9.05 (0.41) | 9.28 (0.15)
  Day 3 | 9.30 (0.61) | 9.37 (0.29) | 9.25 (0.39) | 9.20 (0.34) | 9.35 (0.14) | 9.38 (0.41) | 9.18 (0.17) | 9.40 (0.24) | 9.13 (0.51) | 9.27 (0.18)
  Day 4 | 9.49 (0.25) | 9.38 (0.27) | 9.37 (0.27) | 9.18 (0.64) | 9.27 (0.12) | 9.40 (0.30) | 9.13 (0.22) | 9.23 (0.50) | 8.88 (0.84) | 9.18 (0.13)
  Day 5 | 9.42 (0.36) | 9.38 (0.21) | 9.37 (0.25) | 9.38 (0.24) | 9.32 (0.25) | 9.24 (0.26) | 9.15 (0.18) | 9.55 (0.17) | 9.20 (0.15) | 9.12 (0.19)
  Day 6 | 9.56 (0.26) | 9.45 (0.29) | 9.45 (0.26) | 9.51 (0.20) | 9.35 (0.10) | 9.36 (0.26) | 9.18 (0.15) | 9.35 (0.24) | 9.32 (0.19) | 9.23 (0.12)
  Day 8 | 9.41 (0.31) | 9.45 (0.20) | 9.28 (0.23) | 9.36 (0.44) | 9.23 (0.10) | 9.33 (0.40) | 8.93 (0.28) | 9.30 (0.22) | 9.18 (0.29) | 9.20 (0.37)
  Day 11 | 9.32 (0.29) | 9.38 (0.33) | 9.07 (0.24) | 9.39 (0.25) | 9.30 (0.39) | 9.19 (0.36) | 8.70 (0.75) | 9.30 (0.22) | 9.13 (0.29) | 9.18 (0.26)
  Day 15 | 9.39 (0.26) | 9.60 (0.17) | 9.40 (0.32) | 9.26 (0.21) | 9.22 (0.19) | 9.06 (0.35) | 8.97 (0.18) | 9.33 (0.22) | 9.28 (0.33) | 9.00 (0.36)
  Day 22 | 9.35 (0.33) | 9.53 (0.45) | 9.18 (0.35) | 9.33 (0.32) | 9.22 (0.17) | 9.14 (0.47) | 8.90 (0.23) | 9.48 (0.13) | 9.18 (0.22) | 9.08 (0.15)
  Day 29 | 9.49 (0.32) | 9.58 (0.22) | 9.40 (0.26) | 9.44 (0.37) | 9.20 (0.27) | 9.32 (0.28) | 8.95 (0.19) | 9.38 (0.13) | 9.17 (0.21) | 9.15 (0.23)
  Day 36: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 36 | 9.40 (0.45) |  |  | 9.33 (0.26) | 9.23 (0.30) | 9.00 (0.26) | 9.07 (0.26) | 9.25 (0.30) | 9.18 (0.35) | 9.00 (0.30)
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 43 | 9.33 (0.39) |  |  | 9.32 (0.21) | 9.37 (0.31) | 9.23 (0.36) | 8.90 (0.26) | 9.28 (0.33) | 9.25 (0.25) | 9.15 (0.33)
  Day 50: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 50 | 9.35 (0.26) |  |  | 9.30 (0.41) | 9.03 (0.21) | 9.40 (0.34) | 8.98 (0.19) | 9.33 (0.33) | 9.43 (0.50) | 9.07 (0.23)
  Day 57: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 57 | 9.46 (0.30) |  |  | 9.47 (0.36) | 9.35 (0.29) | 9.18 (0.49) | 9.28 (0.17) | 9.33 (0.29) | 9.25 (0.27) | 9.02 (0.21)
  Day 64: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 64 | 9.22 (0.15) |  |  |  |  | 9.28 (0.42) | 8.90 (0.36) | 9.25 (0.07) |  | 9.18 (0.35)
  Day 71: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 71 | 9.36 (0.18) |  |  |  |  | 9.47 (0.47) | 9.05 (0.36) | 9.20 (0.14) |  | 9.20 (0.14)
  Day 78: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 78 | 9.30 (0.24) |  |  |  |  | 9.31 (0.32) | 9.07 (0.40) | 9.20 (0.00) |  | 9.12 (0.34)
  Day 85: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 85 | 9.12 (0.08) |  |  |  |  | 9.47 (0.35) | 8.82 (0.31) | 9.10 (0.28) |  | 9.05 (0.26)

32. Secondary Outcome: Ionized Calcium Over Time
Time Frame: Day 1 predose and at 4, 6, 8, 10, 12 hours, days 2, 3, 4, 5, 6, 8, 11, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, and 85
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo SC | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Placebo IV | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Number analyzed (Participants) | 14 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
mg/dL
  Day 1 Pre-dose: number analyzed (Participants) | 13 | 6 | 6 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 1 Pre-dose | 5.02 (0.20) | 4.95 (0.18) | 5.02 (0.16) | 5.01 (0.18) | 4.88 (0.08) | 5.07 (0.18) | 4.85 (0.10) | 5.30 (0.12) | 5.18 (0.15) | 5.27 (0.15)
  Day 1 Hour 4 | 5.06 (0.20) | 5.02 (0.17) | 5.10 (0.13) | 5.11 (0.24) | 5.03 (0.10) | 5.12 (0.32) | 4.95 (0.08) | 5.40 (0.14) | 5.35 (0.18) | 5.40 (0.09)
  Day 1 Hour 6 | 4.97 (0.19) | 4.93 (0.10) | 4.98 (0.10) | 4.97 (0.21) | 4.93 (0.08) | 5.06 (0.24) | 4.87 (0.12) | 5.10 (0.14) | 5.28 (0.15) | 5.30 (0.09)
  Day 1 Hour 8 | 4.93 (0.14) | 4.92 (0.15) | 5.00 (0.11) | 5.00 (0.21) | 4.90 (0.06) | 5.04 (0.27) | 4.78 (0.12) | 5.30 (0.08) | 5.28 (0.17) | 5.30 (0.09)
  Day 1 Hour 10 | 5.06 (0.20) | 5.00 (0.09) | 5.05 (0.10) | 5.11 (0.19) | 4.95 (0.15) | 5.07 (0.34) | 4.88 (0.12) | 5.30 (0.12) | 5.32 (0.18) | 5.38 (0.15)
  Day 1 Hour 12 | 5.01 (0.18) | 4.95 (0.08) | 5.00 (0.15) | 5.01 (0.20) | 4.93 (0.16) | 5.03 (0.30) | 4.80 (0.11) | 5.28 (0.22) | 5.25 (0.10) | 5.33 (0.08)
  Day 2 | 5.04 (0.20) | 5.03 (0.16) | 4.92 (0.17) | 5.03 (0.17) | 4.98 (0.12) | 5.04 (0.19) | 4.88 (0.15) | 5.28 (0.10) | 5.08 (0.08) | 5.18 (0.10)
  Day 3 | 5.06 (0.19) | 5.00 (0.13) | 4.97 (0.14) | 5.00 (0.14) | 4.95 (0.08) | 5.12 (0.20) | 4.85 (0.05) | 5.28 (0.13) | 5.17 (0.12) | 5.25 (0.14)
  Day 4 | 5.05 (0.17) | 4.97 (0.15) | 4.85 (0.16) | 5.03 (0.10) | 4.87 (0.12) | 5.11 (0.20) | 4.82 (0.08) | 5.23 (0.17) | 5.20 (0.09) | 5.17 (0.14)
  Day 5 | 5.02 (0.18) | 4.93 (0.10) | 4.88 (0.25) | 5.04 (0.12) | 4.93 (0.12) | 5.04 (0.19) | 4.80 (0.06) | 5.40 (0.14) | 5.18 (0.12) | 5.15 (0.14)
  Day 6 | 5.02 (0.16) | 4.91 (0.14) | 4.97 (0.12) | 5.06 (0.11) | 4.88 (0.10) | 5.02 (0.14) | 4.80 (0.06) | 5.23 (0.10) | 5.23 (0.12) | 5.05 (0.10)
  Day 8 | 5.02 (0.17) | 4.98 (0.08) | 4.92 (0.10) | 5.01 (0.24) | 4.83 (0.10) | 4.89 (0.18) | 5.00 (0.14) | 5.23 (0.17) | 5.17 (0.12) | 5.07 (0.19)
  Day 11 | 5.01 (0.14) | 5.05 (0.14) | 4.93 (0.14) | 5.06 (0.17) | 4.90 (0.13) | 4.92 (0.15) | 5.00 (0.11) | 5.23 (0.13) | 5.20 (0.13) | 5.10 (0.20)
  Day 15 | 5.05 (0.16) | 5.10 (0.19) | 4.92 (0.12) | 5.02 (0.16) | 4.83 (0.12) | 4.98 (0.19) | 5.00 (0.06) | 5.20 (0.22) | 5.25 (0.12) | 5.07 (0.12)
  Day 22 | 5.03 (0.17) | 5.05 (0.18) | 4.82 (0.12) | 4.92 (0.16) | 4.85 (0.08) | 5.08 (0.17) | 5.05 (0.08) | 5.18 (0.24) | 5.12 (0.15) | 5.05 (0.21)
  Day 29 | 5.13 (0.17) | 5.05 (0.08) | 4.92 (0.17) | 5.02 (0.20) | 4.85 (0.08) | 5.22 (0.12) | 5.03 (0.16) | 5.28 (0.17) | 5.22 (0.10) | 5.13 (0.20)
  Day 36: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 36 | 5.16 (0.17) |  |  | 4.96 (0.14) | 5.07 (0.16) | 5.11 (0.18) | 4.96 (0.16) | 5.28 (0.13) | 5.18 (0.10) | 5.18 (0.15)
  Day 43: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 43 | 5.18 (0.23) |  |  | 4.99 (0.15) | 5.22 (0.13) | 5.26 (0.21) | 5.02 (0.08) | 5.23 (0.17) | 5.30 (0.13) | 5.18 (0.12)
  Day 50: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 50 | 5.21 (0.19) |  |  | 5.19 (0.16) | 5.20 (0.11) | 5.16 (0.11) | 5.00 (0.13) | 5.28 (0.15) | 5.32 (0.13) | 5.15 (0.14)
  Day 57: number analyzed (Participants) | 10 | 0 | 0 | 9 | 6 | 9 | 6 | 4 | 6 | 6
  Day 57 | 5.26 (0.14) |  |  | 5.22 (0.14) | 5.22 (0.10) | 5.21 (0.15) | 5.18 (0.13) | 5.33 (0.17) | 5.23 (0.08) | 5.25 (0.15)
  Day 64: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 64 | 5.18 (0.11) |  |  |  |  | 5.22 (0.18) | 5.13 (0.14) | 5.15 (0.07) |  | 5.17 (0.14)
  Day 71: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 71 | 5.18 (0.08) |  |  |  |  | 5.38 (0.16) | 5.12 (0.18) | 5.30 (0.28) |  | 5.20 (0.13)
  Day 78: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 78 | 5.28 (0.08) |  |  |  |  | 5.30 (0.17) | 5.15 (0.19) | 5.15 (0.07) |  | 5.27 (0.15)
  Day 85: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0 | 6
  Day 85 | 5.24 (0.11) |  |  |  |  | 5.36 (0.13) | 5.13 (0.22) | 5.20 (0.14) |  | 5.23 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of treatment up until day 29 for the 0.1 mg/kg and 0.3 mg/kg SC treatment groups, up to 57 days for the 1 mg/kg and 3 mg/kg IV/SC groups and for up to 85 days for the 5 mg/kg and 10 mg/kg SC/IV groups.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo SC | Placebo IV | Romosozumab 0.1 mg/kg SC | Romosozumab 0.3 mg/kg SC | Romosozumab 1.0 mg/kg SC | Romosozumab 10.0 mg/kg SC | Romosozumab 3.0 mg/kg SC | Romosozumab 5.0 mg/kg SC | Romosozumab 1.0 mg/kg IV | Romosozumab 5.0 mg/kg IV
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/4 | 0/6 | 0/6 | 0/9 | 1/6 | 0/6 | 0/9 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 9/14 | 2/4 | 4/6 | 4/6 | 1/9 | 5/6 | 5/6 | 6/9 | 1/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (N=14) | Placebo IV (N=4) | Romosozumab 0.1 mg/kg SC (N=6) | Romosozumab 0.3 mg/kg SC (N=6) | Romosozumab 1.0 mg/kg SC (N=9) | Romosozumab 10.0 mg/kg SC (N=6) | Romosozumab 3.0 mg/kg SC (N=6) | Romosozumab 5.0 mg/kg SC (N=9) | Romosozumab 1.0 mg/kg IV (N=6) | Romosozumab 5.0 mg/kg IV (N=6)
HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (N=14) | Placebo IV (N=4) | Romosozumab 0.1 mg/kg SC (N=6) | Romosozumab 0.3 mg/kg SC (N=6) | Romosozumab 1.0 mg/kg SC (N=9) | Romosozumab 10.0 mg/kg SC (N=6) | Romosozumab 3.0 mg/kg SC (N=6) | Romosozumab 5.0 mg/kg SC (N=9) | Romosozumab 1.0 mg/kg IV (N=6) | Romosozumab 5.0 mg/kg IV (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BASEDOW'S DISEASE (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
AXILLARY PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 2 | 0 | 0
INJECTION SITE HAEMORRHAGE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
INJECTION SITE REACTION (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
THIRST (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HORDEOLUM (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
TINEA PEDIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.